CLINICAL TRIAL: NCT01810692
Title: Cross-sectional Study to Assess the Handling , Patient Satisfaction, and Preference for Inhalation Devices in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Preference Tiotropium Respimat Study in COPD
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.514
Record Dates: First submitted 2013-03-12; First posted 2013-03-13 (Estimated); Results first posted 2015-03-26 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Group 1
  Interventions: Device: Group1:Spiriva® Respimat®
- Group 2
  Interventions: Device: Group2:Hirobriz®/Oslif®/Onbrez® Breezhaler®

INTERVENTIONS:
Device: Group1:Spiriva® Respimat® — COPD patients using Respimat®
  Groups: Group 1
Device: Group2:Hirobriz®/Oslif®/Onbrez® Breezhaler® — COPD patients using Breezhaler®®
  Groups: Group 2

SUMMARY:
In COPD the patient's ability to use inhalers correctly and their preference for the inhaler are both important factors in selecting an appropriate treatment for COPD. This is a cross-sectional study where satisfaction, preference and handling of two different devices such as Respimat and Breezhaler will be evaluated by using the validated PASAPQ in COPD patients

DETAILED DESCRIPTION:
Purpose:

Study Design:

ELIGIBILITY:
Inclusion criteria:

1. All patients must sign an informed consent consistent with International Conference on Harmonization - Good Clinical Practice (ICH-GCP) guidelines prior to participation in the study and conducting any study procedures.
2. Adult male or female patients with chronic obstructive pulmonary disease (COPD) for less than a year who follow usual clinical practice of the participant sites and who are on treatment with Spiriva® Respimat®, Hirobriz® Breezhaler® / Onbrez® Breezhaler® / Oslif® Breezhaler® for at least of 3 months but not more than maximum of 6 months before the informed consent date.

Exclusion criteria:

1. Previously included in this study or currently participating in another interventional study.
2. Visual, cognitive, or motor impairment that as judged by the investigator does not allow the patient to independently read and complete the questionnaire.
3. Patients who are treated simultaneously with both respiratory medications (Spiriva® Respimat® and Hirobriz® Breezhaler® / Onbrez® Breezhaler® / Oslif® Breezhaler®).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COPD
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (15):
- Spain (15):
  - Boehringer Ingelheim Investigational Site 13, A Coruña
  - Boehringer Ingelheim Investigational Site 5, Barcelona
  - Boehringer Ingelheim Investigational Site 6, Barcelona
  - Boehringer Ingelheim Investigational Site 8, Barcelona
  - Boehringer Ingelheim Investigational Site 12, Burgos
  - Boehringer Ingelheim Investigational Site 14, Galdako.
  - Boehringer Ingelheim Investigational Site 11, Laredo
  - Boehringer Ingelheim Investigational Site 1, Málaga
  - Boehringer Ingelheim Investigational Site 3, Mérida
  - Boehringer Ingelheim Investigational Site 15, Palma de Mallorca
  - Boehringer Ingelheim Investigational Site 9, Pozuelo de Alarcón
  - Boehringer Ingelheim Investigational Site 7, Sabadell
  - Boehringer Ingelheim Investigational Site 2, Seville
  - Boehringer Ingelheim Investigational Site 10, Torrelodones
  - Boehringer Ingelheim Investigational Site 4, Villanueva de la Serena

RESULTS

PARTICIPANT FLOW:
Groups:
- Spiriva Respimat: Patients treated with Spiriva Respimat, 2.5 µg, 2 puffs once daily, oral inhalation.
- Hirobriz/Onbrez/Oslif Breezhaler: Patients treated with Hirobriz Breezhaler, Onbrez Breezhaler or Oslif Breezhaler, 150µg / 300µg inhalation powder, once daily oral inhalation.
Period: Overall Study
Arm/Group | Spiriva Respimat | Hirobriz/Onbrez/Oslif Breezhaler
Started | 77 | 77
Completed | 77 | 77
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients from the Treated Set (TS) who reported information about the last prescription of inhalation devices before the start of the study.
Groups:
- Spiriva Respimat: Chronic Obstructive Pulmonary Disease (COPD) patients treated with Spiriva Respimat, 2.5 µg, 2 puffs once daily, oral inhalation.
- Hirobriz/Onbrez/Oslif Breezhaler: Chronic Obstructive Pulmonary Disease (COPD) patients treated with Hirobriz Breezhaler, Onbrez Breezhaler or Oslif Breezhaler, 150µg / 300µg inhalation powder, once daily oral inhalation.
- Total: Total of all reporting groups
Arm/Group | Spiriva Respimat | Hirobriz/Onbrez/Oslif Breezhaler | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.7 (10.0) | 67.0 (9.9) | 68.4 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 69 | 70 | 139
Time since diagnosis of COPD [Mean (Standard Deviation); unit: years] | 6.3 (6.0) | 5.9 (5.4) | 6.1 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Total Mean Score of the Validated Patient Satisfaction and Preference Questionnaire (PASAPQ)
Description: Patient satisfaction with regard to the total score of the handling of the inhaled devices performed by means of a PASAPQ. All questions were answered on a 7-point scale ranging from 1= very dissatisfied to 7 = very satisfied).To calculate the total score, the sum of the 13 items of the two domains (performance and convenience) was transformed to a 0- (least) to 100- (most) point scale which is scaled positively:higher scores represent higher levels of satisfaction.
Time Frame: day 1
Population: Patients from the Full Analysis Set (FAS) which includes all patients from TS who provide evaluable data for the total score of the PASAPQ.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spiriva Respimat | Hirobriz/Onbrez/Oslif Breezhaler
Number analyzed (Participants) | 77 | 77
units on a scale | 80.71 (10.47) | 79.92 (12.68)

2. Secondary Outcome: Total Performance PASAPQ Score.
Description: All questions were answered on a 7-point scale ranging from 1= very dissatisfied to 7 = very satisfied).To calculate the domain scores, the sum of the items of the performance domain was transformed to a 0- (least) to 100- (most) point scale which is scaled positively:higher scores represent higher levels of satisfaction.
Time Frame: day 1
Population: Patients from FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spiriva Respimat | Hirobriz/Onbrez/Oslif Breezhaler
Number analyzed (Participants) | 77 | 77
units on a scale | 82.50 (12.57) | 78.20 (15.84)

3. Secondary Outcome: Total Convenience PASAPQ Score
Description: All questions were answered on a 7-point scale ranging from 1= very dissatisfied to 7 = very satisfied).To calculate the domain scores, the sum of the items of the convenience domain was transformed to a 0- (least) to 100- (most) point scale which is scaled positively:higher scores represent higher levels of satisfaction.
Time Frame: day 1
Population: Patients from FAS.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spiriva Respimat | Hirobriz/Onbrez/Oslif Breezhaler
Number analyzed (Participants) | 77 | 77
units on a scale | 78.62 (11.28) | 81.93 (11.74)

4. Secondary Outcome: Overall Satisfaction Question
Description: The overall satisfaction ranges from 1=very dissatisfied to 7=very satisfied.
Time Frame: day 1
Population: Patients from FAS
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Spiriva Respimat | Hirobriz/Onbrez/Oslif Breezhaler
Number analyzed (Participants) | 77 | 77
units on a scale | 5.96 (0.80) | 5.90 (1.21)

ADVERSE EVENTS:
Time Frame: 1 day
Description: The occurrence of adverse events was assessed from signed informed consent to the completion of the questionnaire.
Arm/Group | Spiriva Respimat | Hirobriz/Onbrez/Oslif Breezhaler
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Other - Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.